CLINICAL TRIAL: NCT03670030
Title: A Pilot Phase 2 Study of Albumin-bound Rapamycin Nanoparticles, ABI-009, in Patients With Metastatic, Unresectable, Low or Intermediate Grade Neuroendocrine Tumors of the Lung or Gastroenteropancreatic System
Brief Title: A Study to testABI-009 in Patients With Metastatic, Unresectable, Low or Intermediate Grade Neuroendocrine Tumors of the Lung or Gastroenteropancreatic System
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Robert Ramirez (Other)
Collaborators: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Robert Ramirez, Principal Investigator, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NET-001
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABI-009 (Experimental): In this study, you will receive ABI-009 given through a vein (intravenous) once weekly for 2 weeks (on days 1 and 8) followed by a week of rest in a 21-day cycle.
  Interventions: Drug: ABI-009

INTERVENTIONS:
Drug: ABI-009 — rapamycin protein-bound nanoparticles for injectable suspension (albumin bound)
  Other Names: nab-rapamycin

SUMMARY:
The purpose of this study is to determine whether ABI-009 will make advanced, malignant neuroendocrine tumor(s) of the lung, gastrointestinal tract and/or pancreas that cannot be removed by surgery smaller and slow the spread of your cancer in patients who have progressed or been intolerant to everolimus. All eligible participants will receive ABI-009, the study drug.

DETAILED DESCRIPTION:
ABI-009, human albumin-bound rapamycin, is an experimental drug. "Experimental" means that the drug has not been approved by the Food and Drug Administration (FDA).

Rapamycin, the active part of the drug, inhibits a biological pathway (mTOR) that certain cancers use to grow. Rapamycin and similar types of drugs have been used in many other tumors, including advanced renal cell carcinoma. A standard mTOR inhibitor used in neuroendocrine tumors is everolimus. The human albumin component of ABI-009 may allow rapamycin to reach cancer cells more effectively.

ABI-009 has not been approved for the treatment of advanced, malignant neuroendocrine tumors of the lung, gastrointestinal tract and/or pancreas. The information from this study might help us identify if ABI-009 is safe and effective in this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable or metastatic patients with typical or atypical carcinoid tumors of the lung or low or intermediate grade gastroenteropancreatic neuroendocrine tumors (GEPNETs).
2. Patients must have measurable disease per RECIST 1.1.
3. Patients must have progressed on everolimus or been intolerant to everolimus.
4. Patients, ≥18 years old, must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
5. Concurrent use of somatostatin analogs (SSAs) is allowed if currently used for symptom control.
6. Adequate liver function:

   1. Total bilirubin ≤1.5 x upper limit of normal (ULN) mg/dL
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (<5 x ULN if the patient has liver metastases).
7. Adequate renal function:

   a. Serum creatinine ≤2 x ULN or creatinine clearance >50 cc/hr (Cockroft-Gault).
8. Adequate biological parameters:

   1. Absolute neutrophil count (ANC) ≥1.5 × 109/L
   2. Platelet count ≥100,000/mm3 (100 × 109/L)
   3. Hemoglobin ≥9 g/dL.
9. Fasting serum triglyceride ≤300 mg/dL; fasting serum cholesterol ≤350 mg/dL.
10. Male or non-pregnant and non-breast feeding female:

    * Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting investigational product (IP) throughout 3 months after last dose of IP and have a negative serum pregnancy test (β-hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. A second form of birth control is required even if she has had a tubal ligation.
    * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after last dose of IP. A second form of birth control is required even if he has undergone a successful vasectomy.
11. Life expectancy of >3 months, as determined by the investigator.
12. Ability to understand and sign informed consent.
13. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients currently undergoing anti-cancer therapy for neuroendocrine tumors (other than SSAs for symptoms).
2. History of allergic reactions to compounds of similar chemical or biologic composition to ABI-009.
3. Known active uncontrolled or symptomatic central nervous system (CNS) metastases. A patient with controlled and asymptomatic CNS metastases may participate in this study. As such, the patient must have completed any prior treatment for CNS metastases ?28 days (including radiotherapy and/or surgery) prior to start of treatment in this study and should not be receiving chronic corticosteroid therapy for the CNS metastases.
4. Active gastrointestinal bleeding.
5. Uncontrolled serious medical or psychiatric illness. Patients with a "currently active" second malignancy other than non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer (staged pathological tumor-2 (pT2) with Gleason Score ≤6 and postoperative prostate-specific antigen (PSA) <0.5 ng/mL), or other adequately treated carcinoma-in-situ are ineligible. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥1 year).
6. Recent infection requiring systemic anti-infective treatment that was completed ≤14 days prior to enrollment (with the exception of uncomplicated urinary tract infection or upper respiratory tract infection).
7. Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy.
8. Unstable coronary artery disease or myocardial infarction during preceding 6 months.
9. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
10. Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfanide) within the 14 days prior to receiving the first dose of ABI-009.
11. Known Human Immunodeficiency Virus (HIV).
12. Known active Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ramirez, DO, Principal Investigator — Ochnser Clinic Foundation
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be made publicly available in the form of poster presentations or journal articles.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABI-009
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ABI-009
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 64 [51 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate at 6 Months Per RECIST v1.1.
Description: Disease control rate at 6 months is the proportion of patients who have partial or complete response or stable disease at 6 months.
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-009
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Percent of Subjects Experiencing Adverse Events
Description: Percent of subjects with >=5% adverse events or grades 3 or 4 adverse events
Time Frame: Continuous from the signing of the informed consent to 28 days after last study treatment, on average 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-009
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Continuous from the signing of the informed consent to 28 days after last study treatment, on average 6 months
Description: Percent of subjects with >=5% adverse events or grades 3 or 4 adverse events
Arm/Group | ABI-009
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-009 (N=5)
Dementia (Nervous system disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-009 (N=5)
Anemia (Blood and lymphatic system disorders) | 3 (21)
Confusion (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 3 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3)
Hypertension (Cardiac disorders) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 3 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Platelet count decrease (Blood and lymphatic system disorders) | 3 (25)
Rash (Skin and subcutaneous tissue disorders) | 3 (13)
Urinary tract infection (Renal and urinary disorders) | 1 (3)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers affecting usefulness interpreting results. Only 2 patients were eligible for analysis of primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT03670030/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03670030/ICF_001.pdf